CLINICAL TRIAL: NCT05047003
Title: Oculogica Portable EyeBOX Study
Acronym: RESTLESS
Status: Completed | Type: Observational
Sponsor: Oculogica, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MTBI003
Record Dates: First submitted 2021-09-10; First posted 2021-09-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Concussion, Brain; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients under evaluation for Suspected Concussion: Device: EyeBOX Model EBX-4 (Portable version)
  Interventions: Diagnostic Test: EyeBOX Model EBX-4 (Portable version)

INTERVENTIONS:
Diagnostic Test: EyeBOX Model EBX-4 (Portable version) — The portable EyeBOX takes less than 4 minutes to complete and involves watching a video move around the perimeter of an LCD monitor positioned in front of the patient while a high-speed camera continuously records gaze positions. The Portable EyeBOX software detects subtle changes in eye movements consistent with concussion and calculates a BOX score.

SUMMARY:
The objective of this study is to assess the accuracy of a portable version of the EyeBOX device, an eye-tracking based diagnostic, in comparison to a clinical reference standard of concussion. The utility of the portable assessment to aid in the monitoring of symptoms over time after an initial diagnosis of concussion will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provide documented informed consent or assent along with guardian consent.
* 2. Have presented, at any time post injury, for any complaint related to an injury involving either a direct force to the head or a blow to the body that has the potential to transmit a rapid acceleration/deceleration of the head, with or without loss of consciousness, with or without external signs of head injury.
* 3. Be 5 to 67 years of age, inclusive.
* 4. Have the ability to provide a complete ophthalmologic, medical, and neurologic history as well as report current medications.

Exclusion Criteria:

* 1. Have penetrating trauma or known skull fracture or intracranial injury.
* 2. Have had a conventional head CT or MRI demonstrating evidence of structural brain injury (subdural, epidural or intraparenchymal hemorrhage, edema/mass effect per attending radiologist read).
* 3. Any of the following conditions, immediately related to the incident injury: loss of consciousness exceeding 30 minutes or best available Glasgow Coma Scale (GCS) score less than 13 within 24 hours or other acute conditions requiring emergency medical management.
* 4. Be blind (no light perception), have missing or non-functional eyes.
* 5. Be unable to open their eyes.
* 6. Have a history of unresolved strabismus, diplopia, amblyopia.
* 7. Have a history of unresolved cranial nerve III, IV, or VI palsy.
* 8. Have a history of unresolved macular edema, retinal degeneration, extensive cataract, or ocular globe disruption.
* 9. Have a history of extensive prior eye surgery or scarring (examples include strabismus surgery, scleral buckle repair of retinal detachment, repair of blow out fractures of the orbit and any procedures that would interfere with extraocular muscle movements; prior cataract surgery or Lasik are not exclusions).
* 10. Have a prior history of unresolved ocular-motor dysfunctions.
* 11. Be intoxicated.

Ages: 5 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive subjects who meet all of the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of initial clinical diagnosis of concussion | Day 0 (when patient first presents for evaluation)
  Sensitivity and Specificity compared to the initial diagnosis of concussion
Diagnostic accuracy of clinical diagnosis of post-concussion symptoms | Up to one year after initial presentation
  Sensitivity and Specificity compared to post-concussion symptoms
Adverse Events | Through study participation, up to one year
  Adverse events occurring during use of the diagnostic device

SECONDARY OUTCOMES:
Diagnostic accuracy to identify increases or decreases in post-concussion symptom severity | Up to one year after initial presentation
  Correlation with increases or decreases in post-concussion symptom severity
Subgroup analyses | Up to one year after initial presentation
  Subgroup analyses will be performed by age, gender, and days since incident injury
Diagnostic accuracy of initial clinical diagnosis of concussion | Day 0 (when patient first presents for evaluation)
  Positive and negative predictive value compared to initial clinical diagnosis of concussion

CONTACTS AND LOCATIONS:
Overall Officials: Rosina Samadani, PhD, Study Director — Oculogica, Inc.; Amy Romandine-Kratz, MD, Principal Investigator — Prevea Health; Mario Chavez, DC, Principal Investigator — Redlands Chiropractic; Brian Lease, PT, Principal Investigator — Westfields Hospital; Yang K Lo, MD, Principal Investigator — CentraCare
Locations (4):
- United States (4):
  - Redlands Chiropractic, Redlands, California
  - CentraCare, Saint Cloud, Minnesota
  - Prevea Health, Green Bay, Wisconsin
  - Westfields Hospital, New Richmond, Wisconsin